CLINICAL TRIAL: NCT01333644
Title: The Role of Inflammation and Aging in HIV-Associated Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: HIV FMD AGING
Record Dates: First submitted 2011-03-01; First posted 2011-04-12 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infection; Cardiovascular Disease; Inflammation
Keywords: HIV Infection; Endothelial function; Cardiovascular Disease; Inflammation; Antiretroviral medication; Treatment naive; Treatment experienced
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, PBMCs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV-Infection: Treated HIV-infected individuals with an undetectable HIV RNA level (< 75 copies RNA/mL, untreated HIV-infected individuals, and HIV-uninfected individuals.

SUMMARY:
It is the central hypothesis of the investigators study that HIV disease is a pro-inflammatory condition, and that years of inflammation result in premature "aging' of the immune system ("immunosenescence"). Just as these changes are thought be causally associated with heart disease in the very old,the investigators postulate that these changes will be associated with early heart disease in the untreated and perhaps treated HIV disease. To address this hypothesis, the investigators will measure immunosenescence in a large cohort of patients who span the entire disease process.

ELIGIBILITY:
Inclusion Criteria:

* HIV controllers: positive for HIV by standard antibody serological determinations with undetectable HIV RNA level (< 75 copies RNA/mL) in absence of therapy
* HIV non-controllers: detectable HIV RNA levels in absence of therapy
* Highly active anti-retroviral therapy responders (HAART responders): on combination antiretroviral therapy with undetectable HIV RNA levels.
* HIV-seronegative participants will also be studied.

Exclusion Criteria:

* Treated individuals that changed antiretroviral regimen within 12 weeks prior to study enrollment.
* Individuals who have started or stopped antihypertensive medication or lipid lowering medication or changed doses of these drugs within 12 weeks of the study will be excluded.
* As nitroglycerin is administered to assess endothelium-independent vasodilation, we also plan to exclude patients who have taken sildenafil, vardenafil, or tadalafil within 72 hours of the endothelial function study, or who are hypotensive (systolic BP <100).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Treated and untreated HIV-infected individuals and HIV-uninfected individuals.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2010-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
brachial artery flow-mediated dilatation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States